CLINICAL TRIAL: NCT00796536
Title: Using fMRI to Evaluate CBT Treatment Response for Patients With Chronic Pain
Brief Title: Using Functional MRI to Evaluate Cognitive Behavioral Therapy Treatment Response in Adults With Chronic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Magdalena Naylor, MD, PhD, Magdalena R. Naylor, MD, PhD, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AR055716 (NIH); R21AR055716 (NIH)
Record Dates: First submitted 2008-11-21; First posted 2008-11-24 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Pain
Keywords: Acute Pain; Low Back Pain; Back Pain; Functional Magnetic Resonance Imaging (fMRI); Cognitive Behavioral Therapy; Pain Education
MeSH Terms: conditions — Chronic Pain; Acute Pain; Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will undergo 12 weeks of group cognitive behavioral therapy (CBT) and a pre- and post-intervention MRI brain scan.
  Interventions: Behavioral: Group cognitive behavioral therapy
- 2 (Active Comparator): Participants will received 12 weeks of pain education and a pre- and post-intervention MRI brain scan.
  Interventions: Behavioral: Pain education

INTERVENTIONS:
Behavioral: Group cognitive behavioral therapy — Each CBT session will last for 90 minutes and will teach participants specific skills to better cope with chronic pain. These skills will include breathing exercises, distraction, and relaxation techniques.
  Arms: 1
Behavioral: Pain education — Patients will receive mailed educational materials to their homes on a weekly basis. Weekly materials will contain information about the nature of chronic back pain, treatment options, exercises and stretching techniques for maintaining strength and flexibility, and proper protection for a healthy back. Pain education is the standard of care for most outpatient clinics.
  Arms: 2

SUMMARY:
Chronic pain is a condition in which pain continues for 1 month or more beyond the usual recovery period for an injury or illness or persists for months or years due to a chronic condition. A commonly used type of psychotherapy called cognitive behavioral therapy (CBT) has been found to be effective in treating people with chronic pain. The purpose of this study is to determine whether and how CBT geared specifically for treating chronic pain can change the way the brain responds to painful emotional and physical stimuli.

DETAILED DESCRIPTION:
Many recent studies have suggested that there is an overlap between pain and emotion-related neurophysiological processes. Several modern pain theories also advocate that pain should be considered as a complex sensory and emotional experience, rather than as an isolated sensory event. In accordance with these theories, it is reasonable to expect that an intervention such as CBT, which teaches patients to understand and control both the emotional and sensory aspects of pain, could alter the brain's responses to both pain and emotionally provocative stimuli and, consequently, change the underlying neural circuitry.

To date, there are no published studies that explore the neurobiological effects of psychotherapeutic approaches, such as CBT, on chronic pain. A previous pilot study showed that the exaggerated amygdala response to negative emotional stimuli in chronic pain patients was normalized after 12 weeks of group CBT, suggesting that CBT may affect at least the emotional component of the pain process. Using functional magnetic resonance imaging (fMRI), which creates a three-dimensional picture of the brain, this study will determine the following: (1) whether CBT treatment changes the function of brain neural circuitry in response to acute noxious physical stimuli and to fearful emotional stimuli; and (2) how altered activation in brain areas associated with the attentional, affective, and sensory aspects of chronic pain relate to measurable improvement in someone's clinical response to group CBT. Directly measuring the effects of CBT on brain function could ultimately improve clinical decision making and contribute to the development of individualized treatment for patients with chronic pain.

Participants will be randomly assigned to receive 12 weeks of either CBT or pain education, which will act as an attention control condition. Each CBT session will last for 90 minutes and will teach participants specific skills to better cope with chronic pain. These skills will include breathing exercises, distraction, and relaxation techniques. Each weekly pain education session, also lasting 90 minutes, will be structured as a group discussion and led by a health care counselor. During the session, participants will receive information about the nature of chronic back pain, talk about treatment options, learn exercises and stretching techniques for maintaining strength and flexibility, and learn how to protect their backs. Every participant will undergo two fMRI examinations: one before treatment and one after treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months of musculoskeletal non-neuropathic pain confined to lumbar or thoracic back
* Meets study threshold for severity of typical pain of 4 or more on a 10-point scale adapted from the McGill Pain Questionnaire
* Has ongoing standard pain management from a physician
* Agrees to participate in this research study

Exclusion Criteria:

* Malignancy
* Reflex sympathetic dystrophy and/or naturopathic pain
* Opioid medication use
* Substance use disorder
* Neurological disorder, such as epilepsy, stroke, or other medical condition that could confound or interfere with the current study
* Major depression or/and dysthymia
* Post traumatic stress disorder or panic disorder
* Left-handedness
* Pregnancy
* History of illicit drug use (cocaine, cannabis, heroin) that can result in altered cognition
* Exceeding the weight limit on the MRI scanner
* Suffering from claustrophobia
* Any of the following: cardiac pacemakers, auto defibrillators, neural stimulators, aneurysm clips, metallic prostheses, cochlear implants, any implanted devices (pumps, infusion devices, stents), permanent eye make-up, intrauterine devices, shrapnel injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Thermal pain threshold, tolerance, perception of acute pain, ability to decrease pain, and brain reactivity | Measured before and after the 12-week intervention

SECONDARY OUTCOMES:
Acute pain perception and brain activation correlated with improvement in clinical outcomes | Measured before and after the 12-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena R. Naylor, MD, PhD, Principal Investigator — MindBody Medicine Clinic, Department of Psychiatry, University of Vermont
Locations (1):
- MindBody Medicine Clinic, Burlington, Vermont, United States

REFERENCES:
- See also: Click here for more information about this study — http://www.med.uvm.edu/mbmc/TB3+CL+BL+3I.asp?SiteAreaID=585